CLINICAL TRIAL: NCT05167656
Title: Intraoral Versus Extraoral Manual Therapy in Subjects With Temporomandibular Disorders. A Randomized Controlled Trial
Brief Title: Intraoral Versus Extraoral Manual Therapy in Subjects With Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Jorge Ballesteros Frutos, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEID/2021/4/087
Record Dates: First submitted 2021-11-22; First posted 2021-12-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers involved in recording outcome measures will not be aware of treatment allocation. Patients will be encouraged to not tell the evaluators about the received treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intraoral Manual Therapy plus exercise and education. (Experimental): Six sessions of intraoral manual therapy plus exercise and counselling.
  Interventions: Other: Intraoral manual therapy; Other: Exercise and counselling
- Extraoral Manual Therapy plus exercise and education. (Experimental): Six sessions of extraoral manual therapy plus exercise and counselling.
  Interventions: Other: Extraoral manual therapy; Other: Exercise and counselling
- Exercise and education. (Active Comparator): Exercise and counselling alone without any manual therapy treatment.
  Interventions: Other: Exercise and counselling

INTERVENTIONS:
Other: Intraoral manual therapy — Six intraoral manual therapy sessions based on ischemic compression and pain pressure release of the temporomandibular region muscles, applied bilateral.
  Arms: Intraoral Manual Therapy plus exercise and education.
Other: Extraoral manual therapy — Six extraoral manual therapy sessions based on ischemic compression, pain pressure release and pressure sliding of the temporomandibular region muscles, applied bilateral.
  Arms: Extraoral Manual Therapy plus exercise and education.
Other: Exercise and counselling — Information about etiology, contributing and related factors, natural history and prognostic of the pathology of temporomandibular disorders.
  Counselling based on: diet, habits like tabacism, stress and anxiety control, physical activity and awareness of dental clenching.
  Exercise daily program based on active and passive mobility of the temporomandibular joint, stretching exercises and self massage.

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effects of intraoral manual therapy versus extraoral manual therapy and compare them with a control group, in the management of patients with temporomandibular disorders regarding pain, strength, quality of life, disability and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral temporomandibular pain for more than one month.
* Older than eighteen.
* No previous treatment to temporomandibular pain in the last 3 months.
* Diagnosed based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

Exclusion Criteria:

* Patients with cervical or cranial trauma or whiplash.
* Diagnosed with systemic disease, like rheumatoid arthritis or fibromyalgia.
* Diagnosed of any vascular or metabolic disease.
* Previous cervical or temporomandibular surgery.
* Dental, medicine or any physical therapy treatment in the last 3 months before the beginning of the interventions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Pain intensity measured with numerical pain rating scale which ranges from 0 points (no pain) to 10 points (worst imaginable pain)

SECONDARY OUTCOMES:
Change in pain pressure threshold | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Pain pressure threshold measured by a digital algometer at several locations of temporomandibular joint.
Change in range of movement of the temporomandibular joint | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Active and passive range of movement measured by a digital caliper.
Change in quality of life | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Quality of life measured with Short Form Health Survey (SF-12). SF-12 ranges from 0 (poor quality of life) to 100 (great quality of life).
Change in disability | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Disability measured with Craniofacial Pain and Disability Inventory (CF-PDI). CF-PDI ranges from 0 (better functional status) to 63 (worse disability).
Change in anxiety | Baseline, change from baseline at 3-week, change from baseline at 6-week, at 1 month after treatment, after 3 months after treatment, after 6 months after treatment.
  Anxiety measured with State-Trait Anxiety Inventory (STAI). STAI ranges from 20 (lower anxiety) to 80 (greater anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No